CLINICAL TRIAL: NCT04049591
Title: A Randomized Trial of Higher vs. Lower Dose Heparin for PCI
Brief Title: Higher vs. Lower Dose Heparin for PCI
Acronym: HD-PCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: HD PCI
Record Dates: First submitted 2019-08-06; First posted 2019-08-08 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Cardiovascular Diseases; Percutaneous Coronary Intervention
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Cluster crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Higher Dose Unfractionated Heparin Treatment Period (Active Comparator): A centre wide policy of administering 100 U/kg bolus of intravenous unfractionated heparin (UFH) for elective percutaneous coronary intervention (PCI) procedures will be implemented during the Higher Dose UFH treatment period.
  Interventions: Drug: Higher Dose UFH
- Lower Dose Unfractionated Heparin Treatment Period (Active Comparator): A centre wide policy of administering 70 U/kg bolus of intravenous UFH for elective PCI procedures will be implemented during the Lower Dose UFH treatment period.
  Interventions: Drug: Lower Dose UFH

INTERVENTIONS:
Drug: Higher Dose UFH — Centre wide policy of administering 100 U/kg bolus of intravenous UFH for elective PCI procedures
  Arms: Higher Dose Unfractionated Heparin Treatment Period
Drug: Lower Dose UFH — Centre wide policy of administering 70 U/kg bolus of intravenous UFH for elective PCI procedures
  Arms: Lower Dose Unfractionated Heparin Treatment Period

SUMMARY:
HD PCI is a multicenter, randomized, registry-based, cluster crossover design trial of higher dose versus lower dose heparin in patients undergoing elective percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
The primary objective of HD PCI is to compare the effect of a policy of higher dose heparin (100 U/kg) use to a policy of lower dose heparin (70 U/kg) use on death, myocardial infarction (MI) or target vessel revascularization (TVR) in patients undergoing elective percutaneous coronary intervention (PCI).

ELIGIBILITY:
Inclusion Criteria:

- Patients undergoing elective PCI

Exclusion Criteria:

* Age <18 years
* Planned chronic total occlusion PCI
* Non-resident precluding follow up through local registries

Hospital (Cluster) Eligibility Criteria

Hospitals will be eligible to participate if they meet the following criteria:

* Submit PCI procedure data to a compatible registry that is able to provide data for the trial
* Site agrees to manage patients as per the higher or lower dose heparin policy in place during the given crossover period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16000 (Estimated)
Dates: Start 2022-03-02 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with any of the following: death, myocardial infarction or target vessel revascularization | up to 30 days after PCI

SECONDARY OUTCOMES:
Number of Participants with major bleeding | up to 30 days after PCI
Number of Participants with any of the following: death, myocardial infarction, target vessel revascularization or major bleeding | up to 30 days after PCI

OTHER OUTCOMES:
Number of Participants with either of the following: death or myocardial infarction | up to 30 days after PCI
Number of Participants with definite stent thrombosis | up to 30 days after PCI

CONTACTS AND LOCATIONS:
Overall Officials: Sanjit Jolly, MD, Principal Investigator — Population Health Research Institute
Locations (1):
- Hamilton Health Sciences, General Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] d'Entremont MA, Lee SF, Wijeysundera HC, Tsang MB, Amlani S, Wassef A, Lavi S, So DYF, Betz J, Tyrwhitt J, Graham J, Cantor WJ, Bagherli A, Vijayaraghavan R, Jolly SS. Design and rationale of the HD PCI trial: A cluster randomized crossover trial of higher vs. lower dose heparin for elective percutaneous coronary intervention. Am Heart J. 2025 Dec 22;294:107330. doi: 10.1016/j.ahj.2025.107330. Online ahead of print. PMID 41443541